CLINICAL TRIAL: NCT03472040
Title: An Open-label Study to Evaluate the Long-term Safety of Daily Oral BCX7353 in Subjects With Type I and II Hereditary Angioedema
Brief Title: A Long Term Safety Study of BCX7353 in Hereditary Angioedema
Acronym: APeX-S
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BCX7353-204
Record Dates: First submitted 2018-02-27; First posted 2018-03-21 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Hereditary Angioedema; HAE; Prophylaxis
Keywords: BCX7353; Hereditary Angioedema; HAE
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BCX7353 150 mg once daily (Experimental)
  Interventions: Drug: BCX7353

INTERVENTIONS:
Drug: BCX7353 — BCX7353 mg oral capsules administered once daily

SUMMARY:
This is an open-label study to evaluate the long term safety and effectiveness of oral treatment with BCX7353 in preventing acute angioedema attacks in patients with Type I and Type II Hereditary Angioedema (HAE).

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with HAE Type I or II who either have participated in a previous BCX7353 study or, in selected countries, in the opinion of the Investigator are expected to derive benefit from an oral treatment for the prevention of angioedema attacks.
* Access to appropriate medication for treatment of acute attacks
* Acceptable effective contraception
* Written informed consent

Key Exclusion Criteria:

* Pregnancy or breast-feeding
* Any clinically significant medical condition or medical history that, in the opinion of the Investigator or Sponsor, would interfere with the subject's safety or ability to participate in the study
* Any laboratory parameter abnormality that, in the opinion of the Investigator, is clinically significant and relevant for this study
* Discontinuation of study drug due to a hypersensitivity reaction BCX7353 in a prior study
* Severe hypersensitivity to multiple medicinal products or severe hypersensitivity/ anaphylaxis with unclear etiology
* Unacceptable noncompliance in a previous BCX7353 study (if applicable) as assessed by the Sponsor or Investigator
* Investigational drug exposure, other than BCX7353, within 30 days prior to the screening visit (or baseline if no screening visit)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 387 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Farkas, MD, Principal Investigator — Semmelweis University, Budapest, Hungary
Locations (87):
- United States (42):
  - Study Center, Birmingham, Alabama
  - Study Center, Scottsdale, Arizona
  - Study Center, Bentonville, Arkansas
  - Study Center, Little Rock, Arkansas
  - Study Center, San Diego, California
  - Study Center, Walnut Creek, California
  - Study Center, Centennial, Colorado
  - Study Center, Colorado Springs, Colorado
  - Study Center, Wheat Ridge, Colorado
  - Study Center, Waterbury, Connecticut
  - Study Center, Tampa, Florida
  - Study Center, Marietta, Georgia
  - Study Center, Normal, Illinois
  - Study Center, Evansville, Indiana
  - Study Center, Indianapolis, Indiana
  - Study Center, Overland Park, Kansas
  - Study Center, Louisville, Kentucky
  - Study Center, Chevy Chase, Maryland
  - Study Center, Boston, Massachusetts
  - Study Center, Ann Arbor, Michigan
  - Study Center, Grand Rapids, Michigan
  - Study Center, Rochester, Minnesota
  - Study Center, Madison, Mississippi
  - Study Center, St Louis, Missouri
  - Study Center, Lincoln, Nebraska
  - Study Center, Charlotte, North Carolina
  - Study Center, Durham, North Carolina
  - Study Center, Cincinnati, Ohio
  - Study Center, Columbus, Ohio
  - Study Center, Clackamas, Oregon
  - Study Center, Happy Valley, Oregon
  - Study Center, Hershey, Pennsylvania
  - Study Center, East Providence, Rhode Island
  - Study Center, Greer, South Carolina
  - Study Center, Austin, Texas
  - Study Center, Dallas, Texas
  - Study Center, Irving, Texas
  - Study Center, San Antonio, Texas
  - Study Center, Murray, Utah
  - Study Center, Seattle, Washington
  - Study Center, Spokane, Washington
  - Study Center, Milwaukee, Wisconsin
- Australia (6):
  - Study Center, Adelaide
  - Study Center, Campbelltown
  - Study Center, Camperdown
  - Study Center, Melbourne
  - Study Center, Murdoch
  - Study Center, Nedlands
- Austria (2):
  - Study Center, Graz
  - Study Center, Vienna
- Study Center, Odense, Denmark
- France (3):
  - Study Center, Grenoble
  - Study Center, Lille
  - Study Center, Paris
- Germany (3):
  - Study Center, Berlin
  - Study Center, Frankfurt
  - Study Center, Ulm
- Study Center, Central, Hong Kong
- Study Center, Budapest, Hungary
- Israel (4):
  - Study Center, Ashkelon
  - Study Center, Haifa
  - Study Center, Tel Aviv
  - Study Center, Tel Litwinsky
- Italy (3):
  - Study Center, Milan
  - Study Center, Padua
  - Study Center, Salerno
- New Zealand (2):
  - Study Center, Auckland
  - Study Center, Wellington
- Study Center, Skopje, North Macedonia
- Study Center, Krakow, Poland
- Serbia (2):
  - Study Center, Belgrade
  - Study Center, Niš
- Study Center, Martin, Slovakia
- Study Center, Cape Town, South Africa
- South Korea (4):
  - Study Center, Daegu
  - Study Center, Donggu
  - Study Center, Gyeonggi-do
  - Study Center, Seoul
- Spain (2):
  - Study Center, Barcelona
  - Study Center, Madrid
- Study Center, Zurich, Switzerland
- United Kingdom (6):
  - Study center, Birmingham
  - Study Center, Bristol
  - Study Center, Cambridge
  - Study Center, London
  - Study Center, Plymouth
  - Study Center, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farkas H, Peter JG, Stobiecki M, Anderson J, Aygoren-Pursun E, Hagin D, Jesenak M, Kessel A, Kiani-Alikhan S, Kinaciyan T, Manning M, Reshef A, Wu A, Iocca HA, Johnston DT, Noble L, Tomita D, Banerji A. Long-term safety and efficacy of once-daily berotralstat in patients with hereditary angioedema: APeX-S final results. Ann Allergy Asthma Immunol. 2025 Sep;135(3):311-319.e6. doi: 10.1016/j.anai.2025.06.004. Epub 2025 Jun 7. PMID 40490218
- [Derived] Peter JG, Desai B, Tomita D, Collis P, Stobiecki M. Assessment of HAE prophylaxis transition from androgen therapy to berotralstat: A subset analysis of the APeX-S trial. World Allergy Organ J. 2023 Nov 6;16(11):100841. doi: 10.1016/j.waojou.2023.100841. eCollection 2023 Nov. PMID 38020288
- [Derived] Riedl MA, Soteres D, Sublett JW, Desai B, Tomita D, Collis P, Bernstein JA; APeX-S Study Investigators. Hereditary angioedema outcomes in US patients switched from injectable long-term prophylactic medication to oral berotralstat. Ann Allergy Asthma Immunol. 2024 Apr;132(4):505-511.e1. doi: 10.1016/j.anai.2023.11.016. Epub 2023 Nov 24. PMID 38006972
- [Derived] Farkas H, Balla Z. A review of berotralstat for the treatment of hereditary angioedema. Expert Rev Clin Immunol. 2023 Feb;19(2):145-153. doi: 10.1080/1744666X.2023.2150611. Epub 2022 Nov 29. PMID 36408587
- [Derived] Riedl MA, Neville D, Cloud B, Desai B, Bernstein JA. Shared decision-making in the management of hereditary angioedema: An analysis of patient and physician perspectives. Allergy Asthma Proc. 2022 Sep 1;43(5):397-405. doi: 10.2500/aap.2022.43.220050. Epub 2022 Jul 12. PMID 35820771
- [Derived] Farkas H, Stobiecki M, Peter J, Kinaciyan T, Maurer M, Aygoren-Pursun E, Kiani-Alikhan S, Wu A, Reshef A, Bygum A, Fain O, Hagin D, Huissoon A, Jesenak M, Lindsay K, Panovska VG, Steiner UC, Zubrinich C, Best JM, Cornpropst M, Dix D, Dobo SM, Iocca HA, Desai B, Murray SC, Nagy E, Sheridan WP. Long-term safety and effectiveness of berotralstat for hereditary angioedema: The open-label APeX-S study. Clin Transl Allergy. 2021 Jun;11(4):e12035. doi: 10.1002/clt2.12035. PMID 34161665

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with a clinical diagnosis of HAE Type 1 or 2 who, in the opinion of the investigator, were expected to benefit from an oral treatment for the prevention of angioedema attacks were considered eligible for the study following assessment of data obtained from screening procedures.
Groups:
- 110 mg Followed by 150 mg Berotralstat: Subjects were initially treated with berotralstat 110 mg per day (QD). Following the results from Part 1 of Study BCX7353-302, all subjects were transitioned to a berotralstat dose of 150 mg QD. Dosing continued for up to 96 weeks (US) / 216 weeks (Rest of World (ROW)).
- 150 mg Berotralstat: Subjects were treated with berotralstat 150 mg QD. Dosing continued for up to 96 weeks (US) / 216 weeks (ROW).
Period: Overall Study
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Started | 100 | 287
Completed | 0 | 1
Not Completed | 100 | 286
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 10 | 23
Not completed — Perceived Lack of Efficacy | 29 | 30
Not completed — Lab Abnormality or Adverse Event (AE) | 7 | 25
Not completed — Intercurrent Illness/Medical Condition | 2 | 3
Not completed — Other - Not Otherwise Specified (NOS) | 4 | 19
Not completed — Subject Non-compliance | 2 | 5
Not completed — Discontinuation due to Rash | 0 | 1
Not completed — Subsequent Ineligibility | 0 | 2
Not completed — Berotralstat Provided by alternative Means (i.e., Early Access Program or Commercially Available) | 46 | 175

BASELINE CHARACTERISTICS:
Groups:
- 110 mg Followed by 150 mg Berotralstat: Subjects were initially treated with berotralstat 110 mg QD. Following the results from Part 1 of Study BCX7353-302, all subjects were transitioned to a berotralstat dose of 150 mg QD. Dosing continued for up to 96 weeks (US) / 216weeks (ROW).
- Total: Total of all reporting groups
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat | Total
Number analyzed (Participants) | 100 | 287 | 387
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 23 | 28
  Between 18 and 65 years | 93 | 253 | 346
  >=65 years | 2 | 11 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.6 (14.04) | 40.5 (15.26) | 39.8 (14.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 180 | 242
  Male | 38 | 107 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 12 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 12 | 12
  White | 82 | 256 | 338
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety & Tolerability
Description: The number and percentage of subjects with treatment-emergent adverse events.
Time Frame: Up to 96 weeks (US) / 216 weeks (Rest of World (ROW)).
Population: The safety population included all subjects who received at least 1 dose of study drug. This population was used in the assessment and reporting of safety data.
Measure: Count of Participants; unit: Participants
Groups:
- 110 mg Followed by 150 mg Berotralstat: Subjects were initially treated with berotralstat 110 mg QD. Following the results from Part 1 of Study BCX7353-302, all subjects were transitioned to a berotralstat dose of 150 mg QD.
- 150 mg Berotralstat: Subjects were treated with berotralstat 150 mg QD.
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Number analyzed (Participants) | 100 | 287
Participants
  TEAE | 94 | 240
  Drug-related TEAE | 58 | 119
  TESAE | 23 | 20
  Drug-related TESAE | 3 | 1
  DMID Grade 3 or 4 TEAE | 18 | 35
  Drug-related DMID Grade 3 or 4 TEAE | 7 | 11
  TEAE leading to study drug discontinuation | 8 | 28
  TEAE leading to study drug interruption | 8 | 32
  Drug-related rash | 5 | 5
  Drug-related rash leading to study drug discontinuation | 1 | 2

2. Secondary Outcome: Incidence of Acute Attacks of Angioedema in Subjects During Treatment
Description: Number of 'adjusted' attacks were assessed. Adjusted attacks included at least 1 symptom of swelling, had a response of 'no' to the diary question, 'In retrospect, could there be an alternative explanation for your symptoms other than an HAE attack (i.e., allergic reaction, viral cold etc.)?', and were considered unique (attack began > 24 hours from the end of the prior attack). Any attack that began within 24 hours from the end of a prior attack was combined with the prior attack.
Time Frame: Up to 96 weeks (US) / 216 weeks (ROW)
Population: The safety population included all subjects who received at least 1 dose of study drug. This population was used in the assessment and reporting of efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Number analyzed (Participants) | 100 | 287
Participants
  Subjects reporting at least 1 attack | 95 | 231
  Subjects reporting at least 1 treated attack | 87 | 214
  Subjects reporting at least 1 untreated attack | 59 | 99

3. Secondary Outcome: The Durability of Response to Treatment
Description: To evaluate if the rate of attacks remains consistent (durable) over time, the monthly attack rate was assessed at 0 to 24 weeks, 24 to 48 weeks, 48 to 96 weeks and 96 weeks until the end of the study. Monthly attack rate was defined as the total number of adjusted HAE attacks experienced during the treatment period adjusted for the length of a month (defined as 28 days) and the number of days the subject was on treatment during that month.
Time Frame: Up to 96 weeks (US) / 216 weeks (ROW)
Population: The safety population included all subjects who received at least 1 dose of study drug. This population was used in the assessment and reporting of efficacy data. The reduced number of subjects analysed at each study period reflects the fact that the maximum duration for US subjects was 96 weeks, as well as subject withdrawal prior to study completion, primarily as a result of Berotralstat being provided by alternative means (i.e., early access program or commercially available).
Measure: Mean (Standard Deviation); unit: HAE attacks per 28 days
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Number analyzed (Participants) | 100 | 287
HAE attacks per 28 days
  0 - 24 weeks | 1.276 (1.2254) | 1.079 (1.4411)
  24 - 48 weeks: number analyzed (Participants) | 77 | 214
  24 - 48 weeks | 1.005 (1.0027) | 0.694 (1.0072)
  48 - 96 weeks: number analyzed (Participants) | 72 | 158
  48 - 96 weeks | 1.121 (1.9573) | 0.591 (0.8217)
  96 weeks - End of Study: number analyzed (Participants) | 58 | 71
  96 weeks - End of Study | 0.770 (1.0394) | 0.725 (0.8395)

4. Secondary Outcome: Patient Reported Quality of Life (QoL) During Treatment
Description: Quality of Life (QoL) specific to hereditary angioedema (HAE) was assessed at baseline and at each study visit until the end of the study. The questionnaire (i.e. AE-QoL) consisted of 17 questions spanning 4 domains (functioning, fatigue/mood, fear/shame, and nutrition). Each AE-QoL question had 5 answer options (scored 1-5), with lower and higher scores indicting less and more adverse impact, respectively. Per-subject scores for each domain were computed using the appropriate scoring algorithm applied to the question response scores for each domain. Per-subject total scores (including all 4 domains) were similarly computed using the question response scores for all 17 questions. The outputs from the scoring algorithm were normalized on a scale ranging from 0 (less adverse impact) to 100 (most adverse impact). The Mean change from baseline (CFB) in AE-QoL total score over time is presented below.
Time Frame: Up to 96 weeks (US) / 216 weeks (ROW)
Population: The safety population was used in the assessment & reporting of efficacy data, & included subjects receiving at least 1 dose of study drug. The reduced number of subjects analysed at each study period reflects that the maximum duration for US subjects was 96 weeks, variation in the number of subjects completing the AE-QoL questionnaire & subject withdrawal prior to study completion, primarily as a result of Berotralstat being provided via an early access program or commercially.
Measure: Mean (Standard Deviation); unit: AE-QoL score - change from baseline
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Number analyzed (Participants) | 81 | 272
AE-QoL score - change from baseline
  Week 4 | -8.85 (18.986) | -10.38 (17.845)
  Week 8: number analyzed (Participants) | 73 | 192
  Week 8 | -11.20 (19.386) | -10.39 (19.690)
  Week 12: number analyzed (Participants) | 70 | 251
  Week 12 | -11.92 (18.484) | -11.47 (18.561)
  Week 24: number analyzed (Participants) | 65 | 224
  Week 24 | -11.58 (17.630) | -11.98 (18.724)
  Week 36: number analyzed (Participants) | 62 | 120
  Week 36 | -11.79 (17.377) | -13.53 (18.556)
  Week 48: number analyzed (Participants) | 62 | 168
  Week 48 | -13.60 (17.339) | -14.08 (19.351)
  Week 60: number analyzed (Participants) | 57 | 113
  Week 60 | -12.81 (15.888) | -16.42 (18.568)
  Week 72: number analyzed (Participants) | 56 | 91
  Week 72 | -13.14 (16.774) | -14.93 (18.991)
  Week 84: number analyzed (Participants) | 52 | 66
  Week 84 | -15.25 (16.776) | -14.70 (17.710)
  Week 96: number analyzed (Participants) | 52 | 74
  Week 96 | -14.72 (15.342) | -17.44 (19.701)
  Week 108: number analyzed (Participants) | 45 | 58
  Week 108 | -14.85 (15.077) | -17.06 (18.963)
  Week 120: number analyzed (Participants) | 43 | 60
  Week 120 | -14.21 (16.140) | -18.20 (18.705)
  Week 132: number analyzed (Participants) | 38 | 55
  Week 132 | -14.58 (15.765) | -16.57 (16.151)
  Week 144: number analyzed (Participants) | 27 | 49
  Week 144 | -13.05 (19.678) | -18.40 (18.081)
  Week 156: number analyzed (Participants) | 26 | 42
  Week 156 | -15.53 (15.823) | -21.29 (20.015)
  Week 168: number analyzed (Participants) | 13 | 20
  Week 168 | -16.70 (13.690) | -22.06 (18.281)
  Week 180: number analyzed (Participants) | 4 | 12
  Week 180 | -21.69 (23.014) | -21.94 (17.652)
  Week 192: number analyzed (Participants) | 1 | 5
  Week 192 | -10.29 (0) | -18.53 (8.860)
  Week 204: number analyzed (Participants) | 0 | 3
  Week 204 |  | -13.24 (11.672)
  Week 216: number analyzed (Participants) | 0 | 2
  Week 216 |  | -17.65 (14.558)

5. Secondary Outcome: Patient's Satisfaction With Medication During Long Term Administration of Berotralstat
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) was completed by subjects at baseline and at each study visit until the end of the study. TSQM scores consisted of 14 items of which 13 items were made up of 3 specific scales (Effectiveness, Side Effects, and Convenience) and 1 global satisfaction scale (Global Satisfaction). At baseline, TSQM questionnaires were completed based on subject's satisfaction with usual medications. At all other time points for collection of TSQM, subjects were asked about their level of satisfaction or dissatisfaction with the study drug. Scale scores were calculated for each scale and were transformed into scores ranging from 0 to 100, with higher scores indicating higher satisfaction. TSQM score and corresponding change from baseline values were calculated at each visit. Note: Subjects in Hong Kong did not complete the TSQM.
Time Frame: Up to 96 weeks (US) / 216 weeks (ROW)
Population: The safety population was used in the assessment & reporting of efficacy data, & included subjects receiving at least 1 dose of study drug. The reduced number of subjects analysed at each study period reflects that the maximum duration for US subjects was 96 weeks, variation in the number of subjects completing the TSQM questionnaire & subject withdrawal prior to study completion, primarily as a result of Berotralstat being provided via an early access program or commercially.
Measure: Mean (Standard Deviation); unit: TSQM score - change from baseline
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
Number analyzed (Participants) | 91 | 277
TSQM score - change from baseline
  Week 4 | -4.1 (35.51) | -1.3 (30.48)
  Week 8: number analyzed (Participants) | 83 | 197
  Week 8 | -0.6 (36.29) | -3.6 (30.38)
  Week 12: number analyzed (Participants) | 78 | 255
  Week 12 | 1.5 (34.35) | -0.1 (31.37)
  Week 24: number analyzed (Participants) | 73 | 227
  Week 24 | 5.4 (34.46) | 1.7 (31.77)
  Week 36: number analyzed (Participants) | 70 | 121
  Week 36 | 5.8 (32.00) | -4.4 (27.41)
  Week 48: number analyzed (Participants) | 70 | 171
  Week 48 | 5.5 (31.79) | 4.1 (27.78)
  Week 60: number analyzed (Participants) | 63 | 115
  Week 60 | 8.0 (30.13) | 3.1 (25.89)
  Week 72: number analyzed (Participants) | 60 | 93
  Week 72 | 9.3 (33.33) | 4.5 (27.32)
  Week 84: number analyzed (Participants) | 55 | 68
  Week 84 | 4.2 (32.32) | 1.3 (20.76)
  Week 96: number analyzed (Participants) | 55 | 76
  Week 96 | 6.2 (35.64) | 5.5 (23.44)
  Week 108: number analyzed (Participants) | 3 | 2
  Week 108 | -7.1 (44.61) | -21.4 (10.10)
  Week 120: number analyzed (Participants) | 47 | 62
  Week 120 | 16.3 (33.06) | 6.8 (22.68)
  Week 132: number analyzed (Participants) | 4 | 5
  Week 132 | 5.4 (41.80) | -5.7 (40.85)
  Week 144: number analyzed (Participants) | 31 | 52
  Week 144 | 18.2 (30.85) | 2.2 (26.82)
  Week 156: number analyzed (Participants) | 9 | 9
  Week 156 | 43.7 (32.23) | -30.2 (32.10)
  Week 168: number analyzed (Participants) | 15 | 20
  Week 168 | -1.4 (22.46) | 6.1 (30.24)
  Week 180: number analyzed (Participants) | 1 | 6
  Week 180 | -7.1 (0) | 11.9 (21.98)
  Week 192: number analyzed (Participants) | 1 | 5
  Week 192 | 0 (0) | 14.3 (8.75)
  Week 204: number analyzed (Participants) | 0 | 1
  Week 204 |  | 14.3 (0)
  Week 216: number analyzed (Participants) | 0 | 2
  Week 216 |  | 10.7 (15.15)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from time of Informed Consent Form signature until the last follow-up visit, approximately 3 weeks following the last dose of study drug; a period of up to 223 weeks in total. Grade 3 and 4 AEs or AEs deemed at least possibly related to use of study drug, were to be followed until the AE resolved or the subject was in a clinically stable condition with regards to the AE.
Groups:
- 110 mg Followed by 150 mg Berotralstat: Subjects were initially treated with berotralstat 110 mg QD. Following the results from Part 1 of Study BCX7353-302, all subjects were transitioned to a berotralstat dose of 150 mg QD. Dosing continued for up to 96 weeks (US) / 216 weeks (ROW).
Arm/Group | 110 mg Followed by 150 mg Berotralstat | 150 mg Berotralstat
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/287
Serious Adverse Events (participants affected / at risk) | 23/100 | 20/287
Other Adverse Events (participants affected / at risk) | 94/100 | 240/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 110 mg Followed by 150 mg Berotralstat (N=100) | 150 mg Berotralstat (N=287)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medical observation (Investigations) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Hereditary angioedema (Congenital, familial and genetic disorders) | 11 (36) | 2 (2)
Splenic hamartoma (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 110 mg Followed by 150 mg Berotralstat (N=100) | 150 mg Berotralstat (N=287)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (19) | 12 (20)
Headache (Nervous system disorders) | 23 (44) | 34 (49)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 42 (51)
Abdominal pain (Gastrointestinal disorders) | 14 (40) | 29 (37)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 14 (16)
Vomiting (Gastrointestinal disorders) | 3 (3) | 17 (17)
Nausea (Gastrointestinal disorders) | 9 (10) | 28 (32)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 18 (25)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 19 (21)
Abdominal discomfort (Gastrointestinal disorders) | 6 (7) | 17 (25)
Nasopharyngitis (Infections and infestations) | 33 (84) | 59 (140)
Upper respiratory tract infection (Infections and infestations) | 14 (31) | 36 (47)
COVID-19 (Infections and infestations) | 10 (10) | 20 (20)
Influenza (Infections and infestations) | 8 (8) | 20 (25)
Urinary tract infection (Infections and infestations) | 7 (10) | 21 (33)
Sinusitis (Infections and infestations) | 10 (20) | 15 (19)
Gastroenteritis (Infections and infestations) | 10 (11) | 12 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT03472040/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/40/NCT03472040/SAP_001.pdf